CLINICAL TRIAL: NCT04754477
Title: A Multicentre, Open, Long-term Clinical Investigation Evaluating Safety, Performance and Patient Reported Outcomes With an Active Osseointegrated Steady-State Implant System in Adult Subjects With Conductive Hearing Loss, Mixed Hearing Loss or Single-sided Sensorineural Deafness.
Brief Title: Long Term Clinical Investigation to Evaluate Clinical Performance, Safety and Patient Reported Outcomes of an Active Osseointegrated Steady-State Implant System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: Statistiska Konsultgruppen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBAS5793
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Results first posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-01

CONDITIONS: Hearing Loss
Keywords: Hearing Loss, Conductive; Hearing Loss, Mixed; Deafness, sensorineural single-sided
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural; Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active Osseointegrated Steady-State Implant System (OSI) (Experimental)
  Interventions: Device: Active Osseointegrated Steady-State Implant System (OSI)

INTERVENTIONS:
Device: Active Osseointegrated Steady-State Implant System (OSI) — System includes the OSI200 implant surgically placed under the skin behind the ear, the BI300 implant osseointegrated in the bone and the external Osia 2 sound process

SUMMARY:
The aim of this clinical investigation is to collect long-term safety and performance data with the Active Osseointegrated Steady-State Implant System by following subjects from the previous Osia clinical investigation CBAS5751. In addition, questions regarding device satisfaction, sound satisfaction, usability and health care utilisation will be asked.

ELIGIBILITY:
Inclusion Criteria:

* Subject has performed Hearing assessment at 3 and/or 6 months in the clinical investigation CBAS5751
* Willing and able to provide written informed consent

Exclusion Criteria:

* Unable to follow investigational procedures, e.g. to complete quality of life scales, or unwilling to comply with the requirements of the clinical investigation as determined by the investigator
* Use of ototoxic drugs that could be harmful to the hearing, as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Ganlöv, MD, Study Director — Cochlear
Locations (3):
- Australia (2):
  - SCIC / NextSense, Gladesville, New South Wales
  - HEARnet Clinical studies, Carlton, Victoria
- Department of Otorhinolaryngology, Head and Neck Surgery Faculty of Medicine. The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request.

REFERENCES:
- [Derived] Cowan R, Lewis AT, Hallberg C, Tong MCF, Birman CS, Ng IH, Briggs R. Clinical performance, safety, and patient-reported outcomes of an active osseointegrated bone-conduction hearing implant system at 24-month follow-up. Eur Arch Otorhinolaryngol. 2024 Feb;281(2):683-691. doi: 10.1007/s00405-023-08133-3. Epub 2023 Aug 8. PMID 37552281

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (20.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Hong Kong | 2
  Australia | 18

OUTCOME MEASURES:

1. Primary Outcome: Number and Type of Reported Adverse Events
Description: The adverse events are collected from the participant's last visit in study CBAS5751 (6 months post-surgery) and categorized by system organ class system
Time Frame: 6 months post-surgery to 24 months post-surgery
Measure: Number; unit: Number of events
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 20
Number of events
  Total number of AEs | 44
  Class congenital, familial and genetic disorders | 1
  Class ear and labyrinth disorders | 16
  Class gastrointestinal disorders | 2
  Class general disorders and administration site conditions | 5
  Class infections and infestations | 3
  Class injury, poisoning and procedural complications | 6
  Class musculoskeletal and connective tissue disorders | 3
  Class neoplasms benign, malignant and unspecified (incl cysts polyps) | 1
  Class nervous system disorders | 1
  Class psychiatric disorders | 3
  Class skin and subcutaneous tissue disorders | 1
  Class surgical and medical procedures | 2

2. Primary Outcome: Number and Type of Reported Device Deficiencies
Description: The device deficiencies are collected from the participant's last visit in study CBAS5751 (6 months post-surgery) and categorized by relationship
Time Frame: 6 months post-surgery to 24 months post-surgery
Measure: Number; unit: Number of events
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 20
Number of events
  Total number of device deficiencies | 19
  Number of deficiencies related to the sound processor | 19

3. Primary Outcome: Concomitant Medication Used
Description: Concomitant medication are collected from the participant's last visit in study CBAS5751 (6 months post-surgery)
Time Frame: 6 months post-surgery to 24 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 19
Participants
  COVID-19 vaccine | 2
  Sofradex for prevention of moist ear | 1
  Otodex for sore or itchy ear | 1
  Soluble aspro clear for bumped head | 1

4. Primary Outcome: Socio-economic Health Care Data Via the Client Service Receipt Inventory (CSRI) Survey
Description: Demographic data (marital status, cohabitation, usual place of residence, education level), employment status, Healthcare utilization and Hearing rehabilitation data are collected
Time Frame: 12 months post-surgery
Population: Data related to ear infection and hearing difficulties are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 19
Participants
  One or more clinical ENT consultation | 8
  Visit to audiologist due to ear infections or hearing difficulties | 8
  One or more diagnostic tests because of ear infections or hearing difficulties | 2
  Stopped, reduced or missed work as a consequence of ear infection and/or hearing difficulties | 0

5. Primary Outcome: Socio-economic Health Care Data Via the Client Service Receipt Inventory (CSRI) Survey
Description: as for outcome 4
Time Frame: 24 months post-surgery
Population: Data related to ear infection and hearing difficulties are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 19
Participants
  One or more clinical ENT consultation | 7
  Visit to audiologist due to ear infections or hearing difficulties | 4
  One or more diagnostic tests because of ear infections or hearing difficulties | 1
  Stopped, reduced or missed work as a consequence of ear infection and/or hearing difficulties | 3

6. Primary Outcome: Change in Audiometric Thresholds With the Active Osseointegrated Steady-State Implant System at 12 Months Post-surgery and 24 Months Post-surgery Compared to Preoperative Thresholds Via an Audiogram
Description: Bone- and air conduction thresholds, masked and unmasked
Time Frame: Baseline before surgery, 12 months and 24 months post-surgery
Population: As per protocol, if failed results regarding Pure Tone Average (PTA4), individual thresholds or Signal to Noise Ratio (SNR) were obtained, both unaided audiograms and BC Direct values could have been used to evaluate if the results depended on impaired unaided hearing or impaired performance of the Osia device. The results were collected, with no failed results for PTA4, individual thresholds or SNR recorded. Therefore the unaided audiograms and BC Direct values were not analysed further.
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in Hearing Performance With the Active Osseointegrated Steady-State Implant System at 12 Months and 24 Months Post-surgery Compared to Last Performed Measurement (3 or 6 Months) in the CBAS5751 Study Assessed Via Audiometric Thresholds
Description: Sound-field (Pure Tone Average 4, mean of 0.5, 1, 2 and 4 kHz)
Time Frame: 3 or 6 months post-surgery, 12 and 24 months post-surgery
Population: Data received for 18 participants.
Measure: Mean (Standard Deviation); unit: dB (decibel)
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 18
dB (decibel)
  From 6 months to 12 months | 2.22 (5.10)
  From 6 months to 24 months | 3.68 (5.15)

8. Secondary Outcome: Change in Hearing Performance With the Active Osseointegrated Steady-State Implant System at 12 and 24 Months Post-surgery Compared to Last Performed Measurement (3 or 6 Months) in the CBAS5751 Study Assessed Via Audiometric Thresholds
Description: Sound-field [0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0 and 8.0 kHz]
Time Frame: 3 or 6 months post-surgery, 12 and 24 months post-surgery
Population: Data were received for 18 participants.
Measure: Mean (Standard Deviation); unit: dB (decibel)
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 18
dB (decibel)
  Change from 6 months to 12 months-250 Hz | 3.33 (8.22)
  Change from 6 months to 12 months-500 Hz | 3.89 (7.78)
  Change from 6 months to 12 months-750 Hz | 2.78 (6.69)
  Change from 6 months to 12 months-1000 Hz | 1.67 (7.28)
  Change from 6 months to 12 months-1500 Hz | 3.89 (6.54)
  Change from 6 months to 12 months-2000 Hz | 0.278 (5.278)
  Change from 6 months to 12 months-3000 Hz | 1.94 (6.67)
  Change from 6 months to 12 months-4000 Hz | 3.06 (5.98)
  Change from 6 months to 12 months-6000 Hz | 3.61 (6.82)
  Change from 6 months to 12 months-8000 Hz | 3.61 (14.33)
  Change from 6 months to 24 months-250 Hz | 4.17 (11.79)
  Change from 6 months to 24 months-500 Hz | 3.89 (6.54)
  Change from 6 months to 24 months-750 Hz | 3.61 (4.47)
  Change from 6 months to 24 months-1000 Hz | 3.89 (7.96)
  Change from 6 months to 24 months-1500 Hz | 5.28 (7.37)
  Change from 6 months to 24 months-2000 Hz | 2.50 (5.49)
  Change from 6 months to 24 months-3000 Hz | 2.78 (7.32)
  Change from 6 months to 24 months-4000 Hz | 4.44 (7.05)
  Change from 6 months to 24 months-6000 Hz | 1.67 (7.07)
  Change from 6 months to 24 months-8000 Hz | 5.00 (11.88)

9. Secondary Outcome: Change in Hearing Performance With the Active Osseointegrated Steady-State Implant System at 12 and 24 Months Post-surgery Compared to Last Performed Measurement (3 or 6 Months) in the CBAS5751 Study Assessed Via Adaptive Speech Recognition in Noise
Description: Speech-to-noise ratio, 50% speech understanding
Time Frame: 3 or 6 months post-surgery, 12 and 24 months post-surgery
Population: Data received for 18 participants.
Measure: Mean (Standard Deviation); unit: db SNR (decibel Speech to Noise Ratio)
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 18
db SNR (decibel Speech to Noise Ratio)
  Change from 6 months to 12 months | -0.106 (2.726)
  Change from 6 months to 24 months | -0.244 (0.913)

10. Secondary Outcome: Change in Hearing Performance With the Active Osseointegrated Steady-State Implant System at 12 and 24 Months Post-surgery Compared to Last Performed Measurement (3 or 6 Months) in the CBAS5751 Study Assessed Via Bone Conduction (BC) Direct
Description: BC direct (0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0 and 6.0 kHz)
Time Frame: 3 or 6 months post-surgery, 12 and 24 months post-surgery
Population: As per protocol, if failed results regarding PTA4, individual thresholds or SNR were obtained, both unaided audiograms and BC Direct values could have been used to evaluate if the results depended on impaired unaided hearing or impaired performance of the Osia device. The results were collected, with no failed results for PTA4, individual thresholds or SNR recorded. Therefore the unaided audiograms and BC Direct values were not analysed further.
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 0

11. Secondary Outcome: Difference in Self-reported Hearing Outcome With the Active Osseointegrated Steady-State Implant System at 12 and 24 Months Post-surgery Compared to Last Performed Measurement (3 or 6 Months) in the CBAS5751 Study
Description: Assessed via Abbreviated Profile of Hearing Aid Benefit (APHAB) questionnaire. APHAB produces a global score and scores for four subscales: Ease of Communication, Reverberation, Background Noise, and Aversiveness. Global score is the average of all subscales. All scales range from 0-100%, where 0% indicates no problem and 100% indicates always problem. A decrease in the APHAB values indicates an improvement. The difference in scores will be presented. A positive value indicates an improvement, a negative value an impairment.
Time Frame: 3 or 6 months post-surgery, 12 and 24 months post-surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 19
units on a scale
  From 6 months to 12 months | -0.067 (7.376)
  From 6 months to 24 months | -0.626 (9.533)

12. Secondary Outcome: Change in Self-reported Hearing Outcome With the Active Osseointegrated Steady-State Implant System at 12 and 24 Months Post-surgery Compared to Last Performed Measurement (3 or 6 Months) in the CBAS5751 Study
Description: Assessed via the Speech, Spatial and Qualities of Hearing Scale (SSQ) questionnaire. Measuring change of speech, spatial and hearing experiences with the Active Osseointegrated Steady-State Implant System. The Total score summarizes the parameters speech, spatial and hearing. A scale from 0 to 10 is used, where 0 represents "can not hear at all", and 10 "hear perfectly". An increase of an SSQ value reflects an improvement. The change in scores will be presented. A positive value indicates improved hearing, a negative value indicates impaired hearing.
Time Frame: 3 or 6 months post-surgery, 12 and 24 months post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 19
score on a scale
  Change from 6 months to 12 months | 0.227 (0.834)
  Change from 6 months to 24 months | -0.155 (1.389)

13. Secondary Outcome: Change in Health-related Quality of Life With the Active Osseointegrated Steady-State Implant System at 12 and 24 Months Post-surgery Compared to Last Performed Measurement (3 or 6 Months) in the CBAS5751 Study
Description: Assessed via the Health Utilities Index (HUI) questionnaire. Change of health status and health related quality of life using the generic quality of life scale Health Utilities Index when wearing the Active Osseointegrated Steady-State Implant System. A health utility value of 1.00 indicates perfect health while a score of 0.00 indicates death. The change in scores will be presented. A positive value indicates an improved quality of life, a negative value indicates impaired quality of life.
Time Frame: 3 or 6 months post-surgery, 12 and 24 months post-surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 19
score on a scale
  Change in comprehensive health status from 6 months to 12 months | 0.006 (0.115)
  Change in vision attribute from 6 months to 12 months | -0.014 (0.085)
  Change in hearing attribute from 6 months to 12 months | 0.024 (0.130)
  Change in speech attribute form 6 months to 12 months | 0.008 (0.069)
  Change in ambulation attribute from 6 months to 12 months | -0.009 (0.039)
  Change in dexterity attribute from 6 months to 12 months | 0.000 (0.000)
  Change in emotion attribute form 6 months to 12 months | -0.009 (0.666)
  Change in cognition attribute from 6 months to 12 months | -0.003 (0.060)
  Change in pain attribute from 6 months to 12 months | 0.015 (0.146)
  Change in comprehensive health status form 6 months to 24 months | -0.045 (0.151)
  Change in vision attribute from 6 months to 24 months | -0.016 (0.086)
  Change in hearing attribute from 6 months to 24 months | 0.003 (0.139)
  Change in speech attribute from 6 months to 24 months | 0.017 (0.080)
  Change in ambulation attribute from 6 months to 24 months | -0.060 (0.163)
  Change in dexterity attribute from 6 months to 24 months | -0.014 (0.062)
  Change in emotion attribute from 6 months to 24 months | -0.005 (0.056)
  Change in cognition attribute from 6 months to 24 months | -0.012 (0.036)
  Change in pain attribute from 6 months to 24 months | -0.001 (0.161)

14. Secondary Outcome: Participant Satisfaction With the Investigational Device (Every-day Situation and Self-esteem) Assessed on a Likert Scale
Description: To express how much they agree or disagree with a particular statement. The scale goes from 1 to 7, where 1 represent Much worse and 7 represent Much better.
Time Frame: 12 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 19
Participants
  Everyday situation-no change | 1
  Everyday situation-a little better | 2
  Everyday situation-somewhat better | 3
  Everyday situation-much better | 13
  Self-esteem-no change | 3
  Self-esteem-a little better | 3
  Self-esteem-somewhat better | 7
  Self-esteem-much better | 6

15. Secondary Outcome: Participant Satisfaction With the Investigational Device (Easiness to Use) Assessed on a Likert Scale
Description: To express how much they agree or disagree with a particular statement. The scale goes from 1 to 5 where 1 represent Very difficult and 5 represent Very easy.
Time Frame: 12 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 19
Participants
  Very easy | 16
  Somewhat easy | 3

16. Secondary Outcome: Participant Satisfaction With the Investigational Device (Durability of the Device and Sound Quality) Assessed on a Likert Scale
Description: To express how much they agree or disagree with a particular statement. The scale goes from 1 to 5, where 1 represent Very dissatisfied and 5 represent Very satisfied.
Time Frame: 12 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 19
Participants
  Durability-neutral | 1
  Durability-satisfied | 9
  Durability-very satisfied | 9
  Sound quality-neutral | 1
  Sound quality-satisfied | 7
  Sound quality-very satisfied | 11

17. Secondary Outcome: Participant Satisfaction With the Investigational Device (Overall Satisfaction) With Question Yes/No.
Time Frame: 12 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 19
Participants
  Yes | 19
  No | 0

18. Secondary Outcome: Participant Satisfaction With the Investigational Device (Every-day Situation and Self-esteem) Assessed on a Likert Scale
Description: as for outcome 14
Time Frame: 24 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 19
Participants
  Every day situation-no change | 0
  Every day situation-a little better | 4
  Every day situation-somewhat better | 3
  Every day situation-much better | 12
  Self-esteem-no change | 2
  self-esteem-a little better | 5
  self-esteem-somewhat better | 5
  self-esteem-much better | 7

19. Secondary Outcome: Participant Satisfaction With the Investigational Device (Easiness to Use) Assessed on a Likert Scale
Description: as for outcome 15
Time Frame: 24 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 19
Participants
  Very easy | 15
  Somewhat easy | 3
  Neither difficult or easy | 1

20. Secondary Outcome: Participant Satisfaction With the Investigational Device (Durability of the Device and Sound Quality) Assessed on a Likert Scale
Description: as for outcome 16
Time Frame: 24 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 19
Participants
  Durability-satisfied | 6
  Durability-very satisfied | 13
  Sound quality-satisfied | 8
  Sound quality-very satisfied | 10
  Sound quality-very dissatisfied | 1

21. Secondary Outcome: Participant Satisfaction With the Investigational Device (Overall Satisfaction) With Question Yes/No.
Time Frame: 24 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 19
Participants
  Yes | 18
  No | 1

22. Secondary Outcome: Daily Use of the Osia 2 Sound Processor at 12 and 24 Months Post-surgery Compared to Last Performed Measurement (3 or 6 Months) in the CBAS5751 Study
Description: Average hours of daily use during the last week before each follow up visit
Time Frame: 3 or 6 months post-surgery, 12 and 24 months post-surgery
Population: Data not collected for all 20 participants at all time points.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 20
hours/day
  At 6 months | 8.25 (4.63)
  At 12 months: number analyzed (Participants) | 19
  At 12 months | 8.74 (3.90)
  At 24 months: number analyzed (Participants) | 19
  At 24 months | 8.47 (5.15)

23. Secondary Outcome: Daily Streaming Time of the Osia 2 Sound Processor at 12 and 24 Months Post-surgery Compared to Last Performed Measurement (3 or 6 Months) in the CBAS5751 Study
Description: Average hours of daily streaming during the last week before each follow up visit
Time Frame: 3 or 6 months post-surgery, 12 and 24 months post-surgery
Population: Data were not received for all 20 participants at all time points.
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 20
hours/day
  At 6 months | 0.400 (0.681)
  At 12 months: number analyzed (Participants) | 19
  At 12 months | 1.16 (2.36)
  At 24 months: number analyzed (Participants) | 19
  At 24 months | 0.789 (1.437)

24. Secondary Outcome: Battery Lifetime of the Osia 2 Sound Processor at 12 and 24 Months Post-surgery Compared to Last Performed Measurement (3 or 6 Months) in the CBAS5751 Study
Description: Average hours of battery lifetime for a single battery during the last week before each follow up visit
Time Frame: 3 or 6 months post-surgery, 12 and 24 months post-surgery
Population: Data not received for all 20 participants at 12 and 24 months.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 20
Hours
  At 6 months | 24.7 (12.9)
  At 12 months: number analyzed (Participants) | 19
  At 12 months | 24.4 (10.3)
  At 24 months: number analyzed (Participants) | 18
  At 24 months | 23.3 (9.2)

25. Secondary Outcome: Magnet Choice of the Osia 2 Sound Processor at 12 and 24 Months Post-surgery Compared to Last Performed Measurement (3 or 6 Months) in the CBAS5751 Study
Description: Magnet strength ranging from 1 to 4, strength 1 being the weakest and 4 the strongest. If the magnet strength has been changed the reason for change is captured in free text
Time Frame: 3 or 6 months post-surgery, 12 and 24 months post-surgery
Population: Data were not received at 24 months for all 20 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 20
Participants
  At 6 months- strength 4 | 9
  At 6 months- strength 3 | 9
  At 6 months- strength 2 | 2
  At 12 months- strength 4 | 8
  At 12 months- strength 3 | 10
  At 12 months- strength 2 | 2
  At 24 months- strength 4: number analyzed (Participants) | 19
  At 24 months- strength 4 | 8
  At 24 months- strength 3: number analyzed (Participants) | 19
  At 24 months- strength 3 | 8
  At 24 months- strength 2: number analyzed (Participants) | 19
  At 24 months- strength 2 | 3

26. Secondary Outcome: Use of SoftWear Pad for the Osia 2 Sound Processor at 12 and 24 Months Post-surgery Compared to Last Performed Measurement (3 or 6 Months) in the CBAS5751 Study
Description: SoftWear pad usage: Yes or No
Time Frame: 3 or 6 months post-surgery, 12 and 24 months post-surgery
Population: Data not received for all 20 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 20
Participants
  At 6 months-Yes | 0
  At 6 months-No | 20
  At 12 months-Yes: number analyzed (Participants) | 19
  At 12 months-Yes | 1
  At 12 months-No: number analyzed (Participants) | 19
  At 12 months-No | 18
  At 24 months-Yes: number analyzed (Participants) | 19
  At 24 months-Yes | 1
  At 24 months-No: number analyzed (Participants) | 19
  At 24 months-No | 18

27. Secondary Outcome: Retention of the Osia 2 Sound Processor at 12 and 24 Months Post-surgery Compared to Last Performed Measurement (3 or 6 Months) in the CBAS5751 Study
Description: Assessed via a Visual Analog Scale (VAS) 100 mm where 0 mm represents insufficient retention and 100 mm excellent retention.
Time Frame: 3 or 6 months post-surgery, 12 and 24 months post-surgery
Population: Data were not received for all 20 participants at all time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 20
units on a scale
  At 6 months | 75.7 (21.9)
  At 12 months: number analyzed (Participants) | 19
  At 12 months | 83.3 (14.2)
  At 24 months: number analyzed (Participants) | 19
  At 24 months | 82.8 (15.0)

28. Secondary Outcome: Wearing Comfort of the Osia 2 Sound Processor at 12 and 24 Months Post-surgery Compared to Last Performed Measurement (3 or 6 Months) in the CBAS5751 Study
Description: Assessed via a Visual Analog Scale (VAS) 100 mm where 0 mm represents no comfort at all and 100 mm excellent comfort.
Time Frame: 3 or 6 months post-surgery, 12 and 24 months post-surgery
Population: Data were not received for all 20 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
Number analyzed (Participants) | 20
units on a scale
  At 6 months | 86.7 (12.4)
  At 12 months: number analyzed (Participants) | 19
  At 12 months | 88.2 (11.0)
  At 24 months: number analyzed (Participants) | 19
  At 24 months | 87.8 (10.3)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Active Osseointegrated Steady-State Implant System (OSI)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Osseointegrated Steady-State Implant System (OSI) (N=20)
Hospitalisation due to unexplained fever (Infections and infestations) | 1 (1)
Hospitalisation for marsupialisation of Bartholin's abscess (Infections and infestations) | 1 (1)
Hospitalisation for bowel surgery for treatment of Hirschsprung's disease (Congenital, familial and genetic disorders) | 1 (1)
Hospitalisation for ankle surgery (Surgical and medical procedures) | 1 (1)
Hospitalisation for hip replacement (Surgical and medical procedures) | 1 (1)
Hospitalisation for surgery to close ileostomy (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Osseointegrated Steady-State Implant System (OSI) (N=20)
Ear infection (Ear and labyrinth disorders) | 4 (8)
Ear pain (Ear and labyrinth disorders) | 2 (4)
Bumped head (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT04754477/Prot_SAP_000.pdf